CLINICAL TRIAL: NCT02297607
Title: Routine Post-Operative Supplemental Nutrition: A Randomized Controlled Trial
Brief Title: Routine Post-Operative Supplemental Nutrition
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor accrual. Patients were reluctant to agree if they would need tube feeding for a month.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Philip W. Carrott, Jr., Assistant Professor of Thoracic Surgery, Medical School, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00091994
Record Dates: First submitted 2014-09-11; First posted 2014-11-21 (Estimated); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer; Esophagectomy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Enteral Nutrition; Osmolite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tube Feeding (Experimental): Study subjects will continue to receive tube feedings (for at least 50% of caloric need) for 1-month post-operatively.
  Interventions: Dietary Supplement: Tube Feeding
- Standard of Care (No Intervention): Tube feeding to continue in the hospital until the patient is taking adequate nutrition by mouth at post-op day #8, or upon discharge,

INTERVENTIONS:
Dietary Supplement: Tube Feeding
  Other Names: Boost; Ensure; Nutren 1.0; Osmolite; Replete
  Arms: Tube Feeding

SUMMARY:
Patients undergoing an esophagectomy will be randomized to receive either (1) routine post-operative tube feeding for 1 month post-operative or (2) usual practice, which is tube feeding to continue in the hospital until the patient is taking adequate nutrition by mouth at POD#8, or upon discharge.

Specific Aim 1 is to determine the occurrence of common complications and readmissions post-operatively between the two patient groups. The investigators hypothesize that routine use of tube feeding may reduce the occurrence of post-operative complications.

Specific Aim 2 is to determine if routine dietary supplementation with enteral tube affects recovery and QOL after esophagectomy. The investigators hypothesize that routine post-operative supplementation will enhance patients recovery and QOL.

For esophagectomy specifically, there is very limited literature evaluating the complication rate and QOL associated with the length of post-operative tube feeding and adequate nutritional requirements. Small randomized studies have not shown a benefit to routine tube feeding, although the numbers were very small, ranging from 12-70 per group. The investigators will randomize 200 patients for the purpose of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an elective esophagectomy
* Jejunal feeding tube placed at the time of surgery

Exclusion Criteria:

* Emergent esophagectomy procedure
* Inability to provide informed consent or to complete testing or data collection
* Unwillingness to be randomized
* Tube feeding dependent on discharge

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Quality of Life after surgery | 6-months post-operatively
  Quality of Life will be assessed using the EORTC QLQ-30 Survey Instrument. Post-operative QOL assessment will be compared to baseline (prior to surgery) QOL assessment.

SECONDARY OUTCOMES:
Jejunostomy tube-specific complications | 2-weeks, 1-month, 3-months and 6-months post-operatively
  j-tube specific complications include infection, bowel obstruction that may require surgical repair, discomfort, diarrhea and dumping syndrome

OTHER OUTCOMES:
Other post-operative complications | 30-days post-operative
  atrial fibrillation, delirium, anastomotic leak, and pneumonia
Costs | 6-months post-operative
  Cost of care
Length of hospital stay | 2-weeks post-operative
  Total length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Philip W Carrott, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

DOCUMENTS (2):
  • Informed Consent Form (2015-10-29): https://cdn.clinicaltrials.gov/large-docs/07/NCT02297607/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2014-06-16): https://cdn.clinicaltrials.gov/large-docs/07/NCT02297607/Prot_SAP_001.pdf